CLINICAL TRIAL: NCT05365607
Title: NightWare Therapeutic Platform for Improving Cardiovascular Health in Adults With Nightmares Associated With PTSD
Brief Title: NightWare and Cardiovascular Health in Adults With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-5027; R21AG075544 (NIH)
Record Dates: First submitted 2022-05-02; First posted 2022-05-09 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Posttraumatic Stress Disorder; Cardiovascular Diseases; Autonomic Dysfunction; Vascular Stiffness; Nightmare; Endothelial Dysfunction
Keywords: sleep; oxidative stress; aging; inflammation; sex/gender
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Cardiovascular Diseases; Primary Dysautonomias; Inflammation

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo (i.e., sham intervention) controlled parallel pilot study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- NightWare (Experimental): In individuals randomized to the active condition, when the stress index is reached during sleep, NightWare will intervene with varying degrees of vibratory stimulation to the watch over a variable length of time to arouse the person out of the nightmare without awaking.
  Interventions: Device: NightWare
- Sham NightWare (Sham Comparator): In individuals randomized to the sham condition, the NightWare intervention will not be enabled.
  Interventions: Device: Sham NightWare

INTERVENTIONS:
Device: NightWare — A wearable digital therapeutic platform consisting of an Apple Watch and iPhone pre-provisioned with Nightware intervention app that will deliver a mild vibration to the watch after detecting individual having a nightmare based on Nightware proprietary algorithm, arousing the individual and disrupting nightmare without awakening.
  Arms: NightWare
Device: Sham NightWare — NightWare device will not deliver an intervention (i.e., no vibration)
  Arms: Sham NightWare

SUMMARY:
The purpose of this study is to determine whether NightWare therapeutic intervention improves biomarkers of vascular aging and autonomic function in adults with nightmares related to PTSD.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is linked to accelerated aging and is associated with increased risk of early-onset cardiovascular disease (CVD) in both men and women. The pathophysiological link between PTSD and CVD is complex and multi-factorial that likely involves premature vascular aging (i.e., large elastic arterial stiffening and vascular endothelial dysfunction) and autonomic dysfunction (e.g., reduced cardiovagal baroreflex sensitivity [cBRS] and heart rate variability [HRV]), along with other mechanisms. Vascular aging and autonomic dysfunction are key antecedents in the development of CVD and individuals with PTSD have greater arterial stiffening, endothelial dysfunction and reductions in cBRS and HRV compared to those without PTSD. The mechanisms by which PTSD contributes to greater vascular and autonomic dysfunction are not completely understood. Sleep is important for cellular and tissue repair, free radical detoxification and reducing oxidative stress and inflammation. Sleep disturbance is a hallmark symptom of PTSD and is associated with biomarkers of vascular aging, autonomic dysfunction and increased risk of CVD. Nightmares, a central feature of PTSD associated-sleep disturbance, are a debilitating symptom that can lead to insomnia or sleep deprivation, daytime sleepiness or fatigue, mood disturbances, cognitive impairments, behavioral problems, or other sequela, that ultimately causes clinically significant distress and impairment in social, occupational and physiological function, as well as increased CVD risk. As such, therapeutic strategies and interventions aimed at reducing nightmare-associated sleep disturbances in individuals with PTSD are clinically important for improving sleep quality, cardiovascular health and risk for future age-associated CVD.

Various psychotherapeutic (e.g., imagery rehearsal therapy [IRT]) and pharmacological (e.g., prazosin) interventions are available for treatment of nightmares associated with PTSD. However, the evidence for their efficacy for addressing sleep disturbances is inconsistent, particularly with pharmaceuticals, and implementation barriers and poor adherence exist with psychotherapy. As such, novel alternative approaches, including the use of digital medicine such as app-based and digital platforms are being developed to improve treatment delivery. NightWare™ digital therapeutic system is one such novel platform that was recently granted Breakthrough Device designation by the FDA for the treatment of nightmares in adults with PTSD. NightWare uses a proprietary application on the Apple Watch® to collect biometric data (i.e., heart rate [HR] and body movement) to learn sleep patterns to create a stress Index. When an individual exceeds this index due to entering a nightmare, NightWare intervenes by sending vibrotactile feedback to the Apple Watch, arousing the individual and interrupting the nightmare without waking or disrupting sleep. Through machine learning, NightWare continually refines its model and knowledge of the person's response, consequently leading to fewer nightmare associated awakenings. In unpublished preliminary studies, NightWare was shown to be safe (no change in suicide risk or daytime sleepiness) and a tendency to have greater improvement in objective measures of sleep quality (i.e., Pittsburgh Sleep Quality Index [PSQI] and amendment for PTSD [PSQI-A]) compared to sham (NightWare but intervention disabled, i.e., no vibration). Whether NightWare improves cardiovascular health in adults with PTSD-related nightmares has yet to be studied.

Accordingly, the investigators are proposing a randomized, double-blind, placebo (i.e., sham intervention) controlled parallel pilot study that will provide the first clinical evidence for the efficacy of the NightWare digital therapeutic system to improve cardiovascular health outcomes in adults with PTSD-related nightmares.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of PTSD via American Psychiatric Association PTSD diagnostic criteria in the fifth edition of its Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
2. Self-report having repetitive nightmares contributing to disrupted sleep
3. age >22 years (rationale is because the device has only been used in adults in 22 years and older);
4. resting blood pressure (BP, <160/100 mmHg);
5. fasted glucose <126 mg/d;
6. non-smokers;
7. no use of vitamin supplements or anti-inflammatory medications, or willing to stop 1 month prior to the vascular visit;
8. Pittsburgh Sleep Quality Index (PSQI) score 6 or higher;
9. Epworth Sleepiness Scale (ESS): Question #8 score above "0" will prompt an additional question: Does individual drive ("get behind the wheel") when they are drowsy? The answer must be "No" to be enrolled in the study due to safety concerns;
10. Wireless Internet and two power outlets where they sleep;
11. Willingness not to use any other application which collects heart rate data on the phone and watch that is used for NightWare.

Exclusion Criteria:

1. uncontrolled hypertension;
2. current or preexisting CVD or cancers (with the exception of past skin cancers) or active infection;
3. diabetes;
4. thyroid dysfunction, defined as an ultrasensitive TSH <0.5 or >5.0 mU/L; volunteers with abnormal TSH values will be re-considered for participation in the study after follow-up evaluation by the PCP with initiation or adjustment of thyroid hormone replacement; or other problems that would interfere with participation in the study;
5. pregnancy or currently breast feeding;
6. current use (or within previous 6 months) of hormone therapy in postmenopausal women;
7. current substance (including marijuana) or alcohol use disorder (past 12 months) per the SCID-5 (see methods of Research Strategy). Adults with past substance or alcohol use disorders will be allowed to participate.
8. Prazosin use; however, participant may be included if tapered by prescribing provider. Taper must be completed and individual must be off prazosin for 2 days prior to enrollment;
9. Participants will be excluded if they report elevated acute risk for suicidal self-directed violence warranting immediate intervention (e.g., suicidal ideation with intent, evaluated by the Columbia-Suicide Severity Rating Scale [C-SSRS]).
10. Current use of varenicline, beta-blockers (unless ophthalmic solutions), or non-dihydropyridines;
11. Shift workers (due to circadian rhythm disruption);
12. Moderate or Severe obstructive sleep apnea (either diagnosed or determined during screening with the WatchPat [AHI≥15];
13. Diagnosis of narcolepsy;
14. Known sleepwalking;

16) Acting out of dreams prior to PTSD trauma; 17) Diagnosis or suspicion of dementia

Ages: 22 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-18 (Actual)

PRIMARY OUTCOMES:
Change in large elastic artery stiffness -carotid artery | Measured before and after 6 weeks of NightWare and sham conditions
  Carotid artery compliance using carotid artery ultrasound
Change in endothelial function | Measured before and after 6 weeks of NightWare and sham conditions
  Brachial artery flow-mediated dilation (FMD) using ultrasound
Change in 1utonomic function - BRS | Measured before and after 6 weeks of NightWare and sham conditions
  Cardiovagal baroreflex sensitivity (cBRS)

SECONDARY OUTCOMES:
Change in large elastic artery stiffness | Measured before and after 6 weeks of NightWare and sham conditions
  Carotid-femoral pulse wave velocity (PWV)
Change in autonomic function - HRV | Measured before and after 6 weeks of NightWare and sham conditions
  Heart rate variability

OTHER OUTCOMES:
Change in PSQI | Measured before and after 6 weeks of NightWare and sham conditions
  sleep questionnaire
Change in PSQI-A | Measured before and after 6 weeks of NightWare and sham conditions
  sleep questionnaire
Change in Epworth sleepiness scale (ESS) | Measured before and after 6 weeks of NightWare and sham conditions
  sleep questionnaire
Change in CESD | Measured before and after 6 weeks of NightWare and sham conditions
  Depression questionnaire
Change in SF-36 | Measured before and after 6 weeks of NightWare and sham conditions
  Perceived psychosocial and health functioning questionnaire
Change in PCL-5 | Measured before and after 6 weeks of NightWare and sham conditions
  Presence and severity of PTSD symptoms questionnaire
Change in Nightmare disorder index | Measured before and after 6 weeks of NightWare and sham conditions
  NDI questionnaire
Change in CSSR-S | Measured before and after 6 weeks of NightWare and sham conditions
  Suicide risk assessment
Change in Norepinephrine | Measured before and after 6 weeks of NightWare and sham conditions
  Marker of sympathetic activity
Change in Oxidized LDL | Measured before and after 6 weeks of NightWare and sham conditions
  Marker of oxidative stress
Change in Total antioxidant status | Measured before and after 6 weeks of NightWare and sham conditions
  Marker of oxidative stress
Change in Interleukin-6 | Measured before and after 6 weeks of NightWare and sham conditions
  Marker of inflammation
Change in C-Reactive Protein | Measured before and after 6 weeks of NightWare and sham conditions
  Marker of inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Kerrie Moreau, PhD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Colorado CCTSI CTRC, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No